CLINICAL TRIAL: NCT03876756
Title: Determination of Risk Factors of Postpartum Urinary Retention: a Retrospective Case-control Study
Brief Title: Determination of Risk Factors of Postpartum Urinary Retention
Acronym: PAUR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 17-020
Record Dates: First submitted 2019-03-06; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Postpartum Acute Urinary Retention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAUR (postpartum acute urinary retention): patients presenting postpartum acute urinary retention.
  Interventions: Other: postpartum acute urinary retention
- Control: patients without postpartum acute urinary retention. This group was selected randomly, respecting a 1:1 matching criteria, including the year of delivery and the age of the patient at delivery.
  Interventions: Other: no postpartum acute urinary retention

INTERVENTIONS:
Other: postpartum acute urinary retention — Collection of risk factors
  Other Names: Collection of risk factors in patients with postpartum acute urinary retention
  Groups: PAUR (postpartum acute urinary retention)
Other: no postpartum acute urinary retention — Collection of risk factors
  Other Names: Collection of risk factors in patients without postpartum acute urinary retention
  Groups: Control

SUMMARY:
Postpartum urinary retention is an uncommon complication of the vaginal delivery. Failure to diagnose it may have a real impact both on the urinary plane but also on the psychological level.

The hypothesis is that the identification of risk factors for the emergence of acute urinary retention would allow preventive management. The investigator conducted a retrospective, comparative, case-control study, including 2 groups of 96 patients who have had a vaginal delivery in the department between 2011 and 2015. The first group included patients with postpartum acute urinary retention (PAUR). The second group, control group, without PAUR, was selected randomly, respecting a 1:1 matching criteria, including the year of delivery and the age of the patient at delivery. The goal was to identify the potential risk factors of post-partum acute urinary retention in order to define a better prevention.

ELIGIBILITY:
Inclusion Criteria:

* vaginal delivery
* between 2011 and 2015
* postpartum acute urinary retention for the first group / without postpartum acute urinary retention for the second group

Exclusion Criteria:

* caesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a vaginal delivery, between 2011 and 2015, in the obstetrics and gynecology department, at the Femme Mère Enfant Hospital, Hospices Civils de Lyon, France.
  The control group, without PAUR, was selected randomly, respecting a 1:1 matching criteria, including the year of delivery and the age of the patient at delivery.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
gestity | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
parity | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with urological antecedents | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with antecedent of PAUR | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
presentation of baby | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
labor duration | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
duration of second stage of labor | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
instrumental delivery | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
dose of local anesthetic for epidural anesthesia | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
duration of epidural anesthesia | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with intact perineum after delivery | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with spontaneous voiding before leaving the delivery room | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with vulvar edema | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)
number of patients with perineal hematoma | between 2011 and 2015
  criteria that may influence the occurrence of postpartum acute urinary retention (risk factors) : criteria related to the patient's history (gestity, parity, urological antecedents, antecedent of PAUR), related to delivery (presentation, labor duration, duration of second stage of labor, instrumental delivery), related to anesthesia (dose of local anesthetic for epidural anesthesia, duration of epidural anesthesia), related to postpartum events (intact perineum after delivery, spontaneous voiding before leaving the delivery room, vulvar edema, perineal hematoma)

CONTACTS AND LOCATIONS:
Overall Officials: Géry LAMBLIN, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No